CLINICAL TRIAL: NCT05514756
Title: VINCI-AD: An Investigation of Transcutaneous Vagus Nerve Stimulation in Mild Cognitive Impairment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tallaght University Hospital (Other)
Responsible Party: Principal Investigator, Sean P Kennelly, Consultant Physician in Geriatric and Stroke Medicine, Director Institute of Memory and Cognition, Associate Professor of Medical Gerontology, Trinity College Dublin, Tallaght University Hospital
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: VINCI-AD
Record Dates: First submitted 2022-07-29; First posted 2022-08-24 (Actual); Last update posted 2024-06-14 (Actual); Status verified 2024-06

CONDITIONS: Mild Cognitive Impairment; Neurocardiogenic Syncope; Memory Impairment; Inflammatory Response; Alzheimer Disease
MeSH Terms: conditions — Cognitive Dysfunction; Syncope, Vasovagal; Memory Disorders; Alzheimer Disease

STUDY DESIGN:
Who Masked: Participant
Masking Description: Participants will be masked to the active vs sham stimulation settings, it is single blinded i.e. study participants are not aware if active or sham stimulation is occurring but the investigator is aware
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Active t-VNS (Active Comparator): Active t-VNS at 8 Hz to the left cymba conchae, acutely for up to 60 minutes
  Interventions: Device: Active t-VNS
- Sham t-VNS (Sham Comparator): Sham t-VNS at 8 Hz to the left earlobe, acutely for up to 60 minutes
  Interventions: Device: Sham t-VNS
- Baseline assessments (Placebo Comparator): Baseline assessments of neurocardiovascular stability, cognition and serum and plasma inflammatory markers per participant serve to act as their own control in this three-part crossover design
  Interventions: Other: Baseline assessments

INTERVENTIONS:
Device: Active t-VNS — Active t-VNS at 8 Hz for up to 60 minutes will be applied to the left cymba conchae
  Arms: Active t-VNS
Device: Sham t-VNS — Sham t-VNS at 8 Hz for up to 60 minutes will be applied to the left earlobe
  Arms: Sham t-VNS
Other: Baseline assessments — Baselines assessments with no stimulation will serve as control in this three-part crossover design
  Arms: Baseline assessments

SUMMARY:
The VINCI-AD study will investigate the impact of non-invasive vagus nerve stimulation (VNS) on memory in participants with existing mild memory impairment. VNS is a safe, existing treatment, licensed in epilepsy and depression. Until recently, stimulating the vagus nerve involved an operation (invasive VNS) but we can now perform VNS by stimulating a nerve in the outer ear with a very gentle current using a small earpiece, called transcutaneous vagus nerve stimulation (t-VNS). Previous studies have indicated that invasive VNS may improve memory in people with no cognitive issues or with dementia. No study has examined the use of t-VNS in people with diagnosed mild memory issues. The main aim of this study is to assess the feasibility of using t-VNS in participants with Mild Cognitive Impairment (MCI). Other objectives include: 1) Determining the optimal stimulation settings to improve memory; 2) Assessment of safety and tolerability of VNS in participants with memory impairment ; 3) Exploration of impact of non-invasive VNS on brain oxygenation via near-infrared spectroscopy (NIRS): 4) Assessment of impact of VNS on blood markers of inflammation: 5) Assessment of impact of VNS on heart rate variability (HRV) and orthostatic stress in participants with memory impairment. The study will enroll participants via the memory assessment service who have been diagnosed with MCI. The study will enroll 40 participants. All eligible participants will undergo three assessments; one as a baseline assessment of neurocardiovascular health, baseline cognitive tests and baseline blood tests. They will then return for two further visits, one while undergoing active stimulation (active t-VNS) and one while undergoing sham stimulation (sham t-VNS).

DETAILED DESCRIPTION:
The VINCI-AD study is an investigator-led, single-centre crossover device study of the NEMOS Cerbomed auricular transcutaneous vagus nerve stimulator (t-VNS) device in participants with diagnosed Mild Cognitive Impairment (MCI). The study will assess the feasibility, safety and tolerability of the study device for the treatment of older adults with MCI. The device contains a small electrode programmed to 8 Hz stimulation, with participant-selected amplitude settings, which delivers a small amount of stimulation to the vagus nerve via the auricular branch of the vagus nerve located in the outer ear. All eligible participants will be enrolled to three visits to the investigation site, wherein they will undergo baseline (no stimulation), active or sham stimulation for 60 minutes during assessments. Participants will act as their own controls with baseline and sham assessments, undertaken 7-10 days apart. The study is single-blinded as the participants will not be aware whether active or sham stimulation is ongoing during respective assessments.

Neurocardiovascular assessments will be initially undertaken at each visit, encompassing heart rate variability (HRV) measures, active stand after minimum of 5 minutes lying supine, with associated near-infrared spectroscopy (NIRS) assessments. Given the orthostatic challenge, each participant will be asked to not consume caffeine prior to assessment and to attend at 14:00 for each assessment. Orthostatic challenges are undertaken indoors at 21 degrees centigrade in the research laboratory.

Cognitive tests undertaken will encompass a computer-based associative memory task, involving 30 Face-Name association pairs; the Sustained Attention Response to Task (SART) test, spatial navigation via Sea Hero Quest Research App and Repeatable Battery for Assessment of Neuropsychological Status examination. NIRS assessment will be ongoing during cognitive testing.

Serum and plasma markers of inflammation including cytokines and chemokines will be taken after each assessment (baseline, active and sham stimulation).

ELIGIBILITY:
Inclusion Criteria:

* Mild Cognitive Impairment as defined by Clinical Dementia Rating Scale Global score of 0.5
* one RBANS index indicating multi-domain amnestic MCI, amnestic MCI or non-amnestic MCI
* native English speakers

Exclusion Criteria:

* significant current depression
* uncorrected vision/hearing loss
* history of brain surgery
* history of epilepsy with seizure event in last year
* taking any pharmacological agents known to significantly increase seizure risk
* arrhythmia including atrial fibrillation
* pacemaker implants
* existing left ear deformity or recent ear trauma
* alcohol dependence
* currently taking DMARDs or immunotherapies

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Safety of acute t-VNS in participants with MCI - assessed via orthostatic challenge | acute (less than 60 minutes)
  Orthostatic stress is measured via the active stand test whereby participants lie supine for 5 minutes with beat to beat blood pressure (BP) monitoring. They then stand and BP response to orthostatic challenge is measured. To standardise assessments, they are all taken at 14:00 each day, without nicotine or caffeine consumed that day, and all routine meds are taken as usual each morning. Orthostatic hypotension is defined by consensus as a sustained reduction of systolic blood pressure (SBP) of at least 20 mmHg or diastolic blood pressure (DBP) of 10 mmHg within 3 minutes of standing
Safety of acute t-VNS in participants with MCI - assessed via structured assessments of adverse events (AEs) and serious adverse events (SAEs) | acute (less than 60 minutes)
  Likert based questionnaires have been developed to assess for the routine side effects noted in the literature for acute t-VNS treatment including pain, skin discomfort, tingling, headache, tinnitus. These Likert scales are rated 1 to 5 with 1 = worse symptoms and 5 = no symptoms, and will be undertaken after active and sham stimulation. Participants will be given contact details of the principal investigator and study coordinator at the hospital who they can contact if they have concerns or any new symptoms arise.
Tolerability of acute t-VNS in participants with MCI | acute (less than 60 minutes)
  Tolerability of the device will be assessed via in-person questionnaires involving Likert-based scales rated 1 to 5 with 1 = poorly tolerable / painful and 5 = no discomfort noted / comfortable

SECONDARY OUTCOMES:
Effect of acute t-VNS on associative memory in participants with MCI | acute (less than 60 minutes)
  The Face Name Association Test is a cross-modal associative memory test involving Face-Name pairs, of which the participant is shown 30 pairs and then asked to recall if they have been shown before, and if so what their name was. t-VNS has been shown to boost associative memory as assessed by this task in cognitively unimpaired older adults, but has not been assessed in those with MCI. Near-infrared spectroscopy (NIRS) assessment will be ongoing during cognitive assessments, and the assessments will be undertaken 3 times, once at baseline, once during sham once during active t-VNS with 7-10 days between assessments
Effect of acute t-VNS on inhibitory control in participants with MCI | acute (less than 60 minutes)
  The Sustained Attention to Response Task (SART) is a computer-based go/no-go task that requires participants to withhold behavioral response to a single, infrequent target (often the digit 3) presented amongst a background of frequent non-targets (0-2, 4-9). There is evidence supporting the role of the SART as a measure of working memory, sustained attention, and impulse/inhibitory control. We will measure participants' response times and accuracy, at baseline, during active and sham t-VNS with near infrared spectroscopy (NIRS) measurements ongoing during task.
Effect of acute t-VNS on spatial navigation in participants with MCI | acute (less than 60 minutes)
  Sea Hero Quest is a multi-platform mobile game designed to help advance the understanding of spatial navigation and 3D navigation, which is one of the first skills lost in dementia. We will measure participants' ability to navigate through 5 pre-specified levels of Sea Hero Quest, specifically speed and accuracy of navigation. Near-infrared specroscopy (NIRS) measurement will be ongoing during assessment and the assessments will be undertaken at baseline, during active and sham t-VNS.
Effect of acute t-VNS on heart rate variability in participants with MCI | acute (less than 60 minutes)
  Heart rate variability (HRV) is an index of the beat- to beat variability between heart beats. Increased vagal tone (and thus vagal action) is generally associated with a lower heart rate and increased HRV. Indices of HRV including SDNN, RMSSD, HF/LF ratio will be obtained during 5 minutes of rest pre -orthostatic stress. Baseline HRV, and HRV during both active t-VNS and sham t-VNS will be obtained for each participant
Effect of acute t-VNS on serum and plasma chemokines and cytokines in participants with MCI | acute (less than 60 minutes)
  Non-invasive VNS has been shown to downregulate inflammatory cytokine release in healthy young participants, but has not been assessed in participants with MCI. We aim to measure a wide array of blood based cytokines and chemokines using the Luminex assay. Serum and plasma samples will be taken at baseline assessment, after acute active t-VNS and sham t-VNS.
Utility of t-VNS device in participants with MCI | acute (less than 60 minutes)
  Participants' objective ability to utilise and troubleshot the t-VNS device will be assessed via modified Kettle test; a brief Occupational Therapy performance-based measure designed to assess cognitive skills in a functional context.

CONTACTS AND LOCATIONS:
Locations (1):
- Tallaght University Hospital, Dublin, Ireland

IPD SHARING:
Plan to Share IPD: No
There is no plan to share individual patient data with other researchers

REFERENCES:
- [Derived] Dolphin H, Dyer AH, Dukelow T, Finucane C, Commins S, Kennelly SP. Safety and feasibility of transcutaneous vagus nerve stimulation in mild cognitive impairment: VINCI-AD study protocol. BMC Neurol. 2023 Aug 2;23(1):289. doi: 10.1186/s12883-023-03320-5. PMID 37532979